CLINICAL TRIAL: NCT05251038
Title: A Phase Ib/II Study of Sotorasib Combined With Chemotherapy for Second Line Treatment of KRAS p. G12C Mutated Advanced Pancreatic Cancer
Brief Title: Study of Sotorasib Combined With Chemotherapy for Second Line Treatment of Pancreas Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funder Decision
Sponsor: Devalingam Mahalingam (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor-Investigator, Devalingam Mahalingam, Sponsor Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCRN GI21-499
Record Dates: First submitted 2022-02-11; First posted 2022-02-22 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-02

CONDITIONS: Pancreatic Cancer; Unresectable Pancreatic Cancer; Metastatic Pancreatic Cancer; KRAS P.G12C
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — sotorasib; irinotecan sucrosofate; Fluorouracil; Leucovorin; Gemcitabine; Taxes; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): Patients will either receive a combination of:
  Sotorasib + Liposomal Irinotecan (nal-IRI) + 5 Fluorouracil (5FU) + Leucovorin (LV)
  OR
  Sotorasib + Gemcitabine (GEM) + Nab-paclitaxel
  *The combination of therapy received is based on the participants prior therapy and of the discretion of their treating physician
  Interventions: Drug: Sotorasib; Drug: Liposomal Irinotecan (nal-IRI); Drug: 5 Fluorouracil (5FU); Drug: Leucovorin (LV); Drug: Gemcitabine (GEM); Drug: Nab paclitaxel

INTERVENTIONS:
Drug: Sotorasib — Intervention instruction outlined in protocol
  Other Names: Lumakras
Drug: Liposomal Irinotecan (nal-IRI) — Intervention instruction outlined in protocol
  Other Names: Onivyde
Drug: 5 Fluorouracil (5FU) — Per standard of care
Drug: Leucovorin (LV) — Per standard of care
Drug: Gemcitabine (GEM) — Per standard of care
Drug: Nab paclitaxel — Per standard of care
  Other Names: Abraxane

SUMMARY:
This is a multicenter, non-randomized, open-label, phase Ib/II study to evaluate the safety, tolerability and efficacy of sotorasib in combination with chemotherapy for patients with advanced KRAS p.G12C mutant pancreatic cancer with progression of disease after first line treatment. There will be a safety lead in to determine the safety and tolerability of the sotorasib in combination with standard chemotherapy. A Simon two-stage design will be employed to evaluate the efficacy of sotorasib in combination with standard of care second line chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

Subject must meet all of the following applicable inclusion criteria to participate in this study:

* Written informed consent and HIPAA authorization for release of personal health information prior to registration. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
* Age ≥ 18 years at the time of consent.
* ECOG Performance Status of 0-1 within 14 days prior to registration.
* Histological or cytological confirmation of pancreatic cancer per AJCC, 8th edition.
* Unresectable or metastatic pancreatic cancer.
* Measurable disease according to RECIST 1.1 within 28 days prior to registration.
* KRAS p. G12C mutation by CLIA certified molecular testing of tumor biopsy or blood based circulating tumor DNA. NOTE: patients must have KRAS p.G12C molecularly confirmed previously or have archived tissue sent for testing and/or undergo biopsy confirming KRAS p.G12C mutation prior to enrollment.
* Demonstrate adequate organ function as defined in the table below. All screening labs to be obtained within 28 days prior to registration:

  * Hematological

    * Absolute Neutrophil Count (ANC): ≥ 1.5 x 109/L
    * Hemoglobin (Hgb): ≥ 9 g/dL; Transfusion permitted within 1 week
    * Platelet Count (Plt): ≥ 100 x 109/L
  * Renal

    * Calculated creatinine clearance1: ≥ 50 mL/min
    * Creatinine (Cr): ≤ 1.5 × upper limit of normal (ULN)
  * Hepatic

    * Bilirubin: ≤ 1.5 × upper limit of normal (ULN)
    * Aspartate aminotransferase (AST) : ≤ 2.5 × ULN; if liver metastases are present, ≤ 5 x ULN
    * Alanine aminotransferase (ALT): ≤ 2.5 × ULN; if liver metastases are present, ≤ 5 x ULN
  * Coagulation ---International Normalized Ratio (INR) or Prothrombin Time (PT) or Activated Partial Thromboplastin Time (aPTT): ≤ 1.5 × ULN; this would not apply to patient's on anti-coagulation therapy (which is permitted on study; EXCEPT Warfarin)
* Progression of disease after first line chemotherapy or recurrent disease either during or < 6 months after last dose of systemic therapy administered for curative intent.
* Prior cancer treatment (including investigational agents) must be completed at least 2 weeks prior to registration and the subject must have recovered from all reversible acute toxic effects of the regimen (other than alopecia or neuropathy) to Grade ≤ 1 or baseline.
* Life expectancy > 3 months in the opinion of the investigator.
* Therapeutic or palliative radiation >/= 2 weeks from registration is allowed provided subject has recovered from all reversible acute toxic effects to Grade </= 1 or baseline.
* Ability to take oral medications.
* Females of childbearing potential with a male partner able to father a child must have a negative pregnancy test within 7 days prior to registration. See protocol for definition of childbearing potential.
* Females of childbearing potential with a male partner able to father a child and male participants able to father a child who have a female partner of childbearing potential must be willing to abstain from heterosexual intercourse or to use effective method(s) of contraception as outlined in protocol.
* As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study.

Exclusion Criteria:

Subjects meeting any of the criteria below may not participate in the study:

* Receipt of two or more lines of chemotherapy. NOTE: Adjuvant or neoadjuvant therapy would be counted as one line of therapy if recurrence or development of metastatic disease occurred within 6 months of last dose of adjuvant/neoadjuvant therapy.
* Previous treatment with a KRASG12C inhibitor.
* Patient unable to receive nal-IRI/5FU/LV or GEM/nab-paclitaxel as second line chemotherapy for pancreatic cancer.
* Grade 2 or higher neuropathy preventing treatment with abraxane containing regimen.
* History of pneumonitis and/or interstitial lung disease (ILD).
* Active brain metastases and/or carcinomatous meningitis from non-brain tumors. NOTE: Subjects who have had brain metastases resected or have received radiation therapy ending at least 4 weeks prior to study Day 1 are eligible if they meet all of the following criteria: a) residual neurological symptoms grade ≤ 2; b) on stable doses of dexamethasone, if applicable; and c) follow-up magnetic resonance imaging (MRI) performed within 28 days shows no new lesions appearing.
* Active infection requiring antibiotics within 1 week of enrollment.
* Cardiac dysfunction:

  * Myocardial Infarction within 6 months of enrollment
  * NYHA > class II CHF
  * unstable angina
  * arrhythmia requiring medication
  * QTc > 470msec.
* Has a known history of Hepatitis B or C. NOTE: Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA. NOTE: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
* Has a known history of Human Immunodeficiency Virus (HIV) infection. NOTE: Subjects with HIV/AIDS with adequate antiviral therapy to control viral load would be allowed if they are stable and have been on treatment for ≥ 4 weeks prior to first dose of study drug(s). Subjects with viral hepatitis with controlled viral load would be allowed while on suppressive antiviral therapy. Testing not required.no testing for HIV is required unless mandated by local health authority.
* Patients with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen, per treating physician discretion, are not eligible for this trial.
* History or presence of hematological malignancies unless curatively treated with no evidence of disease ≥ 2 years.
* Surgery within 28 days of enrollment.
* Known dihydropyrimidine dehydrogenase deficiency.
* Use of known CYP3A4 and P-gp sensitive substrates (with a narrow therapeutic window), within 14 days or 5 half-lives of the drug or its major active metabolite, whichever is longer, prior to study Day 1 that was not reviewed and approved by the principal investigator.
* Use of strong inducers of CYP3A4 (including herbal supplements such as St. John's wort) within 14 days or 5 half-lives (whichever is longer) prior to study day 1 that was not reviewed and approved by the principal investigator.
* Female subjects who are breastfeeding or who plan to breastfeed while on study and through the timeframe as described in protocol (NOTE: breast milk cannot be stored for future use while the mother is being treated on study). Male participants who plan to donate sperm while on study and through the timeframe as described in protocol.
* Use of warfarin. NOTE: use of low molecular weight heparin (LMWH) are permitted.
* Acid reducing agents including proton pump inhibitors (PPIs) and H2 receptor antagonists. Alternative agents to acid reducing agents are permitted. If an acid-reducing agent cannot be avoided, administer sotorasib 4 hours before or 10 hours after acid-reducing agent use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 2 years
  Clinical activity will be assessed by overall response rate (ORR). ORR is defined as the percentage of patients whose best response is Complete Response (CR) plus those with Partial Response (PR) based on RECIST 1.1.

SECONDARY OUTCOMES:
Assess Adverse Events | 2 months
  Characterize the safety and tolerability of patients receiving sotorasib combined with chemotherapy for second line treatment of pancreas cancer. Determine safety and tolerability as determined by NCI CTCAE v 5.0
Progression Free Survival (PFS) | 6 months, 1 year, and 2 years
  Determine progression free survival (PFS) including the 6- month, 1- year, 2-year and median progression free survival. PFS is defined from the date from first dose of study drug administration (C1D1) until the date of first documentation of progressive disease by RECIST 1.1 or death from any cause, whichever comes first
Duration of Response (DoR) | 2 years
  Determine the Duration of Response (DOR). DOR is defined from the date of first documentation of response to treatment, to the date of first documentation of progressive disease by RECIST 1.1 or death, whichever comes first, in patients who experience a response.
Disease Control Rate (DCR) | 2 years
  Determine the Disease Control Rate (DCR). DCR is defined as the percentage of patients whose best response is complete response (CR) plus partial response (PR) plus stable disease (SD) by RECIST 1.1.
Overall Survival (OS) | 2 years
  Determine Overall Survival (OS). OS is assessed from the date of registration to the study until the date of death from any cause for up to 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Devalingam Mahalingam, MD, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No